CLINICAL TRIAL: NCT04243681
Title: Combination of Autologous Mesenchymal and Hematopoietic Stem Cell Infusion in Patients With Decompensated Cirrhosis: A Pilot Study
Brief Title: Combination of Autologous MSC and HSC Infusion in Patients With Decompensated Cirrhosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECR/346/Inst/AP/2013
Record Dates: First submitted 2019-08-14; First posted 2020-01-28 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-01

CONDITIONS: Cirrhosis, Liver
Keywords: Mesenchymal Stem Cell; Hematopoetic Stem cell; Autologous transfusion
MeSH Terms: conditions — Liver Cirrhosis | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination MSC and HSC (Experimental): Patient will receive a combination of mesenchymal and Hematopoetic stem cell through hepatic artery under fluroscopic guidance
  Interventions: Combination Product: CD 34 and MSC infusion
- Standard of care for Cirrhosis management (Active Comparator): Diuretics, Hepatoprotective agents and Lactulose
  Interventions: Drug: Standard of care for Cirrhosis management

INTERVENTIONS:
Combination Product: CD 34 and MSC infusion — Combination of stem cells
  Other Names: Stem cell infusion
  Arms: Combination MSC and HSC
Drug: Standard of care for Cirrhosis management — Drugs used for Cirrhosis management such as Diuretics, Hepatoprotective agents and Lactulose
  Arms: Standard of care for Cirrhosis management

SUMMARY:
Though the results of autologous CD34+ cell infusion and MSC in independent studies have shown promise, yet they are yet to reach the desired long term outcome. The possible postulation for this is possibly because when using autologous CD34+ cell infusion, the inflammatory milieu of the liver may not be conducive for sustained effects of the mobilized CD 34+ cells. MSC have immunomodulatory effect (ref) and may improve the liver environment making it more beneficial for the CD34+ cells to function and survive. In addition, MSC has ben shown to produce hepatocyte growth factor which is protective against liver injury and beneficial for liver regeneration (shown in above tables). However, it remains to be understood how MSCs promote liver stem stem cells to differentiate into hepatocytes or expand the residual hepatocyte population. MSC can also directly inhibit the activation of hepatic stellate cells, the main source of extracellular matrix via MSC derived IL 10 and TNF-αand may also induce hepatic stellate cell apoptosis. Current lacunae in cell based therapy is based on the poor consensus and understanding on the best type of cells to be used, the ideal number of cells, the most appropriate route of administration and the need for repeat dosing . The concept that combination of autologous hematopoietic and mesenchymal stem cells infusion may be more beneficial than infusing any one of them alone has been discussed in many scientific forums but there are no study till date to either see the safety as well as the efficacy of this proof of concept .

With this above background data, we propose a study design which will be a safety study for combination use of autologous CD34+ and MSC

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-70 years
* Clinically diagnosed for hepatic cirrhosis having a Child Pugh score of B or MELD >10 but below 20
* Not willing for immediate liver transplantation either due to lack of donor tissue or financial issues
* Platelet count of > 80,000 and INR <1.6
* Life expectancy of at least 3 months based on MELD score and Child Pugh Score
* Ability to give informed consent

Exclusion Criteria:

* Age less than 20 or more than 70 years
* Have liver tumors or history of any other cancer
* Pregnant or lactating women
* Patients with hepato-renal syndrome and acute kidney injury (Any creatinine > 1.6 will be excluded)
* Evidence of ongoing sepsis - as per Surviving sepsis guideline
* Recent gastrointestinal bleeding or spontaneous bacterial peritonitis (within last one month)
* Any HIV positive patients
* Co-morbid conditions such as severe cardiac and/or pulmonary disease
* Inability to give informed consent

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
To assess the safety of combination of hematopoetic and mesenchymal stem cell in patients of liver cirrhosis. | Up to 6 months
  Any adverse events after the use of combination stem cell treatment would be recorded:
  * Bone marrow aspiration related complications such as pain (>6 on VAS) and bleeding from the site.
  * Leukapheresis related complications such as hypotension and hypocalcemia.
  * Hepatic artery catheterization related complications such as pain or discomfort at the catheter insertion site, bleeding and infection.
  * Post MSC and CD34 infusion related adverse reactions would be recorded using CDSCO form.

SECONDARY OUTCOMES:
Change in MELD (Model for End stage Liver disease) score. | Up to 6 months
  Difference in MELD score from baseline to follow-up period.
Change in Child Pugh score. | Up to 6 months
  Difference in Child Pugh score from baseline to follow-up period.
Change in the percentage of CD 34 cells in liver. | Up to 6 months
  To assess improvement in the percentage of CD 34 cells in liver by performing a paired liver biopsy- before and after infusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Asian Institute Of Gastroenterology, Hyderabad, Telangana, India

REFERENCES:
- [Background] Amer ME, El-Sayed SZ, El-Kheir WA, Gabr H, Gomaa AA, El-Noomani N, Hegazy M. Clinical and laboratory evaluation of patients with end-stage liver cell failure injected with bone marrow-derived hepatocyte-like cells. Eur J Gastroenterol Hepatol. 2011 Oct;23(10):936-41. doi: 10.1097/MEG.0b013e3283488b00. PMID 21900788
- [Background] Hang HL, Xia Q. Role of BMSCs in liver regeneration and metastasis after hepatectomy. World J Gastroenterol. 2014 Jan 7;20(1):126-32. doi: 10.3748/wjg.v20.i1.126. PMID 24415865
- [Background] Gordon MY, Levicar N, Pai M, Bachellier P, Dimarakis I, Al-Allaf F, M'Hamdi H, Thalji T, Welsh JP, Marley SB, Davies J, Dazzi F, Marelli-Berg F, Tait P, Playford R, Jiao L, Jensen S, Nicholls JP, Ayav A, Nohandani M, Farzaneh F, Gaken J, Dodge R, Alison M, Apperley JF, Lechler R, Habib NA. Characterization and clinical application of human CD34+ stem/progenitor cell populations mobilized into the blood by granulocyte colony-stimulating factor. Stem Cells. 2006 Jul;24(7):1822-30. doi: 10.1634/stemcells.2005-0629. Epub 2006 Mar 23. PMID 16556705
- [Derived] Sharma M, Pondugala PK, Jaggaihgari S, Mitnala S, Krishna VV, Jaishetwar G, Naik P, Kumar P, Kulkarni A, Gupta R, Singh JR, Darisetty S, Sekharan A, Reddy DN, Rao GV, Syeda F, Jagtap N, Rao PN. Safety Assessment of Autologous Stem Cell Combination Therapy in Patients With Decompensated Liver Cirrhosis: A Pilot Study. J Clin Exp Hepatol. 2022 Jan-Feb;12(1):80-88. doi: 10.1016/j.jceh.2021.03.010. Epub 2021 Apr 2. PMID 35068788